CLINICAL TRIAL: NCT04466137
Title: A Multi-centers, Randomized, Open-labeled, Positive-controlled, Phase 3 Study to Evaluate the Safety and Efficacy of YPEG-rhG-CSF, Once-per-cycle, in Patients With Malignancies Receiving Myelosuppressive Chemotherapy.
Brief Title: Phase 3 Study to Evaluate the Safety and Efficacy of YPEG-rhG-CSF in Malignancies Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB1801CSF
Record Dates: First submitted 2020-06-29; First posted 2020-07-10 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Non-Myeloid Malignancy
Keywords: G-CSF; Human Granulocyte Colony-Stimulating Factor; Febrile Neutropenia; Neutropenia; Myelosuppressive Chemotherapy; FN
MeSH Terms: conditions — Febrile Neutropenia; Neutropenia | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- YPEG-rhG-CSF 2mg (Experimental): YPEG-rhG-CSF 2mg
  Interventions: Drug: YPEG-rhG-CSF
- YPEG-rhG-CSF 33μg/kg (Experimental): YPEG-rhG-CSF 33μg/kg
  Interventions: Drug: YPEG-rhG-CSF
- Positive Control Group (Active Comparator): rhG-CSF/PEG-rhG-CSF
  Interventions: Drug: rhG-CSF/PEG-rhG-CSF

INTERVENTIONS:
Drug: YPEG-rhG-CSF — YPEG-rhG-CSF 2mg, single s.c. at day 3 of each cycles, up to 4 cycles. 21 day one cycles.
  Arms: YPEG-rhG-CSF 2mg
Drug: YPEG-rhG-CSF — YPEG-rhG-CSF 33μg/kg, single s.c. at day 3 of each cycles, up to 4 cycles. 21 day one cycles.
  Arms: YPEG-rhG-CSF 33μg/kg
Drug: rhG-CSF/PEG-rhG-CSF — rhG-CSF 5μg/kg/day, s.c. from day 3 to day 14 or until neutrophils recover to exceed 5.0×10^9 cells/L, whichever comes first, in the first cycle. Patient can still continue rhG-CSF 5μg/kg/day, or covert to PEG-rhG-CSF 6mg/Cycle in the following 2-4 cycle. 21 day one cycles.
  Arms: Positive Control Group

SUMMARY:
This phase 3 study is aimed to evaluate the safety and efficacy of YPEG-rhG-CSF in reducing the infection manifested by febrile neutropenia in patients with non-myeloid malignancy who receiving Myelosuppressive Chemotherapy which is likely to cause clinically significant febrile neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology and/or cytology diagnosed as breast cancer (BC) or non-small cell lung cancer (NSCLC), and patients with breast cancer is suitable to receive TAC(Docetaxel,Doxorubicin combined with Cyclophosphamide) chemotherapy, while patients with NSCLC is suitable to receive DC(Docetaxel combined with Carboplatin) chemotherapy.
* Age ≥18 yrs.
* Weight ≥45 kg.
* Karnofsky Score ≥ 70.
* Life Expectancy ≥ 3 months.
* Peripheral blood test: WBC≥3.5×10^9 cells/L, PLT≥100×10^9 cells/L. ANC≥1.5×10^9 cells/L.
* Understand and voluntarily sign the informed consent form.

Exclusion Criteria:

* Receiving chemotherapy within two months prior to screening.
* Previously or plan to receive radiotherapy (>25% total bone marrow volume).
* Evidence of tumor metastasis in bone marrow.
* Lack of awareness.
* Uncontrolled infection or using of antibiotics within 72hrs prior to screening.
* Previously received or plan to undergoing bone marrow or organ transplants.
* Patients with bleeding tendency, e.g. prolonged prothrombin time of more than 3 seconds.
* Dysfunction in heart,lung, liver, kidney, or other major organs or systems; ALT>2.5 ULN (upper limit of normal), TBil >2.5 ULN (ALT>2.5 ULN, total bilirubin >2.5 ULN for patients with liver metastasis), HBsAg positive, anti-HCV positive, evidence of liver decompensation, or Cr >1.5 ULN.
* Pregnant or lactating females.
* Malignancy other than BC or NSCLC.
* Hypersensitivity to rhG-CSF or any component of the investigational Products.
* Subject enrolled in any other studies within 3 months prior to screening.
* Drug abuser or alcoholics.
* Any other conditions which in the opinion of the investigator precluded enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Mean Duration of Severe Neutropenia (DSN) During Cycle 1. | At the end of Cycle 1 (21 days one cycle)
  Mean duration of severe neutropenia, defined as number of consecutive days with absolute neutrophil count (ANC) <0.5 × 10^9 cells/l (grade 4 neutropenia)

SECONDARY OUTCOMES:
Incidence of Febrile neutropenia(FN). | Cycle1 to Cycle 4(21 days one cycle)
  FN defines as the ANC counts is less than < 0.5 × 10^9 cells/L or ANC counts between 0.5 × 10^9 cells/L and 1.0 × 10^9 cells/L but probably to decline to less than 0.5×10^9 cells/L within 48hrs, and body temperature is higher than 38.3 degrees Celsius or higher than 38.0 degrees Celsius and lasting for more than 1hr.
Mean duration of DSN. | Cycle2 to Cycle 4 (21 days one cycle)
Incidence of Grade 3 neutropenia. | Cycle1 to Cycle 4 ( 21 days one cycle)
  Grade 3 neutropenia defines as the ANC count is less than 1.0×10^9 cells/L.
Mean duration of grade 3 neutropenia. | Cycle1 to Cycle 4(21 days one cycle)
Neutrophils dynamic changes from baseline. | Cycle1 to Cycle 4 ( 21 days one cycle)
Time of neutrophils recovering to over 2.0×10^9 cells/L after nadir. | Cycle1 to Cycle 4 (21 days one cycle)
Proportion of patients with antibiotic usage. | Cycle1 to Cycle 4 ( 21 days one cycle)
Proportion of patients experienced infection. | Cycle1 to Cycle 4 ( 21 days one cycle)
Proportion of patients fulfilling expected chemotherapy. | Cycle1 to Cycle 4 (21 days one cycle)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Shi Y, Wang X, Pei Z, Shi H, Zhang Y, Yi T, Mei J, Guo Y, Dong Y, Ma T, Zhang Q, Jia X, Zhu Z, Xu S, Liu Y, Niu H, Jiang W, Jiang X, Zhou S, Sun L. Telpegfilgrastim for chemotherapy-induced neutropenia in patients with non-small cell lung cancer: a multicentre, randomized, phase 3 study. BMC Cancer. 2025 Mar 17;25(1):490. doi: 10.1186/s12885-025-13736-6. PMID 40098083